CLINICAL TRIAL: NCT06318286
Title: First-line Pembrolizumab Plus Platinum Doublet Chemotherapy With Lenvatinib in Unresectable Malignant Pleural Mesothelioma：Multi-Institutional, Single-Arm Phase 2 Trial
Brief Title: Study of Pembrolizumab Plus Chemotherapy With Lenvatinib for Malignant Pleural Mesothelioma
Acronym: PENINSULA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hyogo Medical University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Prof. Kozo Kuribayashi, MD PhD, Professor, Hyogo Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK3475-IIT-60977
Record Dates: First submitted 2024-02-27; First posted 2024-03-19 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Pembrolizumab; Lenvatinib
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — lenvatinib; Pemetrexed; Cisplatin; Carboplatin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label study to evaluate the efficacy and safety of lenvatinib in combination with pembrolizumab and chemotherapy in patients with malignant pleural mesothelioma. Patients 18 years of age or older will be eligible for enrollment if they had histologically confirmed unresectable malignant pleural mesothelioma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lenvatinib, Pemetrexed, Cisplatin/Carboplatin, and Pembrolizumab (Experimental): In induction treatment, study interventions include oral lenvatinib, 8 mg quaque die (QD), and pembrolizumab, 200 mg, carboplatin (AUC 5 mg/mL/min) or cisplatin (75 mg/m2), and pemetrexed, 500 mg/m2 all given by intravenous (IV) infusion on Day 1 of a 21-day cycle. Lenvatinib, pembrolizumab, carboplatin/cisplatin, and pemetrexed combination treatment will be given for 4-6 cycles, after which participants may receive maintenance treatment with Lenvatinib, 20 mg QD, and pembrolizumab, 200 mg. Lenvatinib and Pembrolizumab may be given for up to a total of 35 cycles.
  Interventions: Drug: Lenvatinib; Drug: Pemetrexed; Drug: Cisplatin/Carboplatin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lenvatinib — Induction treatment: lenvatinib, 8 mg QD on Day 1 of a 21-day cycle for 4-6 cycles. Maintenance treatment: Lenvatinib, 20 mg QD may be given for up to a total of 35 cycles.
  Other Names: E7080
Drug: Pemetrexed — Pemetrexed, 500 mg/m2 will be given by intravenous (IV) infusion on Day 1 of a 21-day cycle for 4-6 cycles.
Drug: Cisplatin/Carboplatin — Carboplatin (AUC 5 mg/mL/min) or Cisplatin (75 mg/m2) will be given by IV infusion on Day 1 of a 21-day cycle for 4-6 cycles.
Drug: Pembrolizumab — Pembrolizumab, 200 mg will be given by IV infusion on Day 1 of a 21-day cycle for up to a total of 35 cycles.
  Other Names: MK-3475

SUMMARY:
In this Phase-II study, the investigators will investigate the efficacy and safety of lenvatinib in combination with pembrolizumab and chemotherapy in patients with malignant pleural mesothelioma.

DETAILED DESCRIPTION:
This is a single-arm, open-label study to evaluate the efficacy and safety of lenvatinib in combination with pembrolizumab and chemotherapy in patients with malignant pleural mesothelioma. The study will consist of a screening phase, a treatment phase, and a follow-up phase. Patients who meet the Inclusion Criteria, do not meet the Exclusion Criteria, and are judged by the investigator to be eligible for this clinical trial will be included. Subjects who meet all of the criteria listed in Criteria for Administration of Investigational Drugs may continue to receive the investigational drug. If a subject receiving investigational drugs meets any of the criteria listed in Discontinuation Criteria of Investigational Drugs, the subject will be evaluated at the end of the treatment phase (at the time of discontinuation) and moved to the post-observation phase.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable advanced or metastatic malignant pleural mesothelioma without prior treatment for malignant pleural mesothelioma
2. Patients expected to survive more than 90 days
3. Patients with a transcutaneous oxygen saturation of 94% or greater measured with a pulse oximeter at rest without oxygen inhalation within 7 days prior to enrollment
4. Patients who have given written consent to participate in this clinical trial (consent by a surrogate is also acceptable, if applicable).
5. Patients who are judged by the principal investigator or coinvestigator to have one or more measurable lesions as defined in Modified RECIST by CT or MRI imaging within 28 days prior to enrollment. However, if the measurable lesion is a pleural lesion only and there is a history of pleurodesis (patients who underwent pleurodesis within 14 days prior to enrollment or pleurodesis with Picibanil within 28 days prior to enrollment are excluded), only patients whose measurable lesion was confirmed on imaging after pleurodesis are eligible.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
7. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of malignant pleural mesothelioma will be enrolled in this study.
8. Have adequate organ function as defined in the following table. All clinical laboratory tests in the screening period should be performed within 10 days prior to the start of study intervention.

Exclusion Criteria:

1. Patients with concomitant or pre-existing severe hypersensitivity reactions to other drugs, including antibody preparations
2. A women of childbearing potential who has a positive urine pregnancy test within 72 hours prior to trial registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
3. Has received prior therapy with an anti-PD-1 (anti-programmed cell death protein 1), anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX40, CD137).
4. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to trial registration.

   Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible Note: If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
5. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
9. Has known active central nervous system metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV) infection.
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg]reactive or HBV-DNA detected) or known active Hepatitis C virus (defined as HCV RNA [qualitative] detected or HCV antibody reactive, if HCV-RNA is not the local SOC) infection.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breast feeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
19. Has had an allogenic tissue/solid organ transplant.
20. Patients with diverticulitis or symptomatic gastrointestinal ulcer disease
21. Patients with pleural effusions requiring drainage more frequently than once every 2 weeks
22. Patients with pericardial or ascites effusions requiring treatment
23. Patients with uncontrolled tumor-related pain
24. Patients with a history of transient ischemic attack, cerebral vascular attack, thrombosis or thromboembolism (pulmonary artery embolism or deep vein thrombosis) within 180 days prior to registration Patients with the following unmanageable or serious cardiovascular diseases

    * Myocardial infarction within 180 days prior to enrollment
    * Uncontrolled angina pectoris within 180 days prior to enrollment
    * New York Heart Association（NYHA）Classification of Cardiac Function Classification III or IV congestive heart failure
    * Uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg for >24 hours) despite appropriate therapy
    * Uncontrolled arrhythmia
25. Patients receiving anticoagulation therapy (excluding antiplatelet therapy including low-dose aspirin) or with diseases requiring such therapy
26. Patients with uncontrolled diabetes mellitus
27. Patients undergoing surgical treatment with local or surface anesthesia within 14 days prior to enrollment
28. Patients undergoing surgical treatment involving general anesthesia within 28 days prior to enrollment
29. Patients who underwent pleurodesis within 14 days prior to enrollment
30. Patients who underwent pleurodesis with picibanil within 28 days prior to enrollment
31. Patients who underwent pericardial adhesion within 28 days prior to enrollment
32. Patients who underwent peritoneal adhesions
33. Patients who received radiation therapy for pain relief within 14 days prior to enrollment
34. Patients who have received radiopharmaceuticals (excluding the use of radiopharmaceuticals for laboratory and diagnostic purposes) within 56 days prior to enrollment
35. Patients who have received other unapproved drugs (including approved drugs not indicated for malignant pleural mesothelioma, drugs administered through clinical studies or unapproved combination drugs, or new formulations) within 28 days (90 days for antibody products) prior to enrollment
36. Patients with prolonged QT interval (QTc, corrected by Fridericia's formula) > 480 msec
37. Participants with proteinuria >1+ on urine dipstick testing/urinalysis will undergo24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥1 g/24 hours will be ineligible.
38. Active hemoptysis (bright red blood ≥ 1/2 teaspoon) or other uncontrolled bleeding within 14 days prior to the study registration.
39. Radiographic evidence of intratumoral cavitations, encasement, or invasion of a major blood vessel. Additionally, the degree of proximity to major blood vessels should be considered because for exclusion because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis after lenvatinib therapy. (In the chest, major blood vessels include the main pulmonary artery, the left and right pulmonary arteries, the 4 major pulmonary veins, the superior or inferior vena cava, and the aorta).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Tumor shrinkage (response rate) (Physician Judgment by Medical Institution, Modified RECIST [Response Evaluation Criteria in Solid Tumors] criteria) | 2 years
  The overall response and the best overall response are the result of the diagnostic imaging evaluated based on Modified RECIST criteria, and the result of the diagnostic imaging does not include clinical progression. The diagnostic imaging for which the overall response is determined other than inevaluable (NE) are considered as the evaluable diagnostic imaging. The response rate is defined as the proportion of participants who have complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression-Free survival (PFS) (Physician Judgment by Medical Institution, Modified RECIST criteria) | 2 years
  Progression-Free survival (PFS) is defined as the time from the date of treatment start to the date of the first documentation of progressive disease (PD), as determined by the overall response of Modified RECIST criteria, or death from any cause, whichever is earlier.
Overall survival time (OS) | 2 years
  Overall Survival time (OS) is defined as the time from the date of treatment start to the date of death from any cause. The Participant without documented death at the last date of confirmation of survival or who is lost to follow-up will be censored at last date of confirmation of survival.
Tumor shrinkage (disease control rate) (Physician Judgment by Medical Institution, Modified RECIST criteria) | 2 years
  The response rate is defined as the proportion of participants who have CR, PR, or stable disease (SD).
Duration of response (Physician Judgment by Medical Institution, Modified RECIST criteria) | 2 years
  The duration of response (DOR) is defined as the time from the first documented evidence of confirmed CR or PR to the first documentation of PD or death due to any cause (whichever is earlier), for participants who demonstrate a confirmed CR or PR.
Best overall response (Physician Judgment by Medical Institution, Modified RECIST criteria) | 2 years
  The best overall response is the result of the diagnostic imaging evaluated based on Modified RECIST criteria, and the result of the diagnostic imaging does not include clinical progression. The diagnostic imaging for which the overall response is determined other than inevaluable (NE) are considered as the evaluable diagnostic imaging.
Incidence of adverse events | 2 years
  Safety, as defined by the rate of any adverse events as assessed by the Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v.5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Kozo Kuribayashi, MD, PhD, Principal Investigator — Department of Respiratory Medicine and Hematology, Hyogo Medical University Hospital
Locations (1):
- Hyogo Medical University Hospital, Nishinomiya, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: No